CLINICAL TRIAL: NCT06925724
Title: A Phase 2 Study of Ivonescimab (Bispecific Antibody Against PD1 and VEGF) For the Treatment of Endometrial (EC) and Cervical (CC) Cancers
Brief Title: A Study of Ivonescimab in People With Endometrial and Cervical Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-007
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer; Cervical Cancer
Keywords: Ivonescimab; 25-007
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm, open-label, single-institution phase II trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivonescimab in People With Endometrial Cancer (Experimental): Study treatment will be given sequentially on the first day of each cycle in a 3-week dosing cycle: Ivonescimab will be administered as 20 mg/kg IV (a fixed dose of 3200 mg for ivonescimab should be used for patients ≥ 160 kg), Q3W administered for 60 minutes (± 10 minutes). The total duration of ivonescimab treatment is up to 24 months.
  Interventions: Drug: Ivonescimab
- Ivonescimab in People With Cervical Cancer (Experimental): Study treatment will be given sequentially on the first day of each cycle in a 3-week dosing cycle: Ivonescimab will be administered as 20 mg/kg IV (a fixed dose of 3200 mg for ivonescimab should be used for patients ≥ 160 kg), Q3W administered for 60 minutes (± 10 minutes). The total duration of ivonescimab treatment is up to 24 months.
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab will be administered as 20 mg/kg IV (a fixed dose of 3200 mg for ivonescimab should be used for patients ≥ 160 kg), Q3W administered for 60 minutes (± 10 minutes)

SUMMARY:
The researchers are doing this study to find out if ivonescimab is an effective treatment for people with endometrial cancer (EC) and/or cervical cancer (CC). The researchers will also look at whether the study drug is safe and causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic/recurrent endometrial or cervical cancer that has progressed after treatment with at least one platinum-based regimen.

  1. Endometrial cancer histologies can include: endometrioid, serous, clear cell, dedifferentiated/undifferentiated, mixed epithelial, adenocarcinoma NOS, and carcinosarcoma.
  2. Cervical cancer histologies can include: squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma
* Measurable disease per RECIST v 1.1 criteria
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
* All patients must have received at least 1 line of platinum-based therapy. Prior PD1 or VEGF therapy is allowed.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤160/90 mmHg.
* Have adequate laboratory values as defined in the following table:
* Hematologic

  * Absolute neutrophil count (ANC) ≥1500/mm3 (≥1.5 × 103/µL)
  * Platelets ≥100,000/µL
  * Hemoglobin ≥9.0 g/dL
  * International Normalized Ratio (INR) ≤1.5
* Renal

  * Creatinine clearance (CrCL) Urinalysis Creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula
  * Urinalysis Urine protein < 2+ (or 24 hour urine protein quantification < 1.0 g)
* Hepatic

  * Total bilirubin ≤1.5 ×ULN (patients with known Gilbert's disease who have bilirubin level ≤ 3 x ULN may be enrolled)
  * AST and ALT ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
  * TSH TSH within normal limits. If TSH is not within normal range despite no symptoms of thyroid dysfunction, normal free T4 level is required.
  * Coagulation Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy, or prophylactic coagulation
* Age ≥18 years at the time of informed consent.
* Patients with treated brain metastases are eligible if follow-up brain imaging after CNS directed therapy shows no evidence of progression. Patients with treated brain metastasis should be excluded if they have any evidence of bleeding, or if they have large lesions at risk of bleeding ie >1.5cm. Patients should also be off corticosteroids at the time of enrollment. Patients with untreated brain metastasis are excluded.
* Not Pregnant and Not Nursing. If with childbearing potential, should have a negative urine pregnancy test at the time of screening.
* Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 90 days after the last dose of the ivonescimab.
* Must have clinical IMPACT data available, if data is not available, must have adequate tissue to available for clinical IMPACT. Patient will consent to 12-245 at enrollment if not previously completed.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Major surgical procedures or serious trauma within 4 weeks prior to enrollment or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to enrollment.
* Patient not recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to enrollment, including but not limited to:

  1. Gastrointestinal bleeding
  2. Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots) Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  3. Nasal bleeding /epistaxis (bloody nasal discharge is allowed)
  4. Need for new therapeutic anticoagulant therapy within 14 days prior to enrollment.

Note: Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to randomization is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.

* History of major diseases before enrollment, specifically:

  1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or vascular disease that required hospitalization within 12 months prior to enrollment, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  2. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before enrollment.
  3. History of arterial thromboembolic event, venous thromboembolic event, , transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to enrollment.
  4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before enrollment
  5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to enrollmen
* Imaging during the screening period shows that the patient has:

  1. Radiologically documented evidence of major blood vessel invasion or encasement by cancer
  2. Radiographic evidence of intratumor cavitation
* Has participated in a study of an investigational agent and received cancer directed study therapy within 4 weeks prior to start of study treatment
* Prolongation of QTc interval (Fredericia) to >480 msec
* Active/Acute Hepatitis B infection

  a. Note: Patients with chronic HBV infection with active disease who meet the criteria for anti HBV therapy should require the patient be on a suppressive antiviral therapy prior to initiation of cancer therapy.
* Active/Acute Hepatitis C infection

  a. Note: Patients who are HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution should be eligible.
* Known intolerance to either of the study drugs (or any of the excipients)
* History of organ allograft (subject has had an allogenic tissue/solid organ transplant)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids (up to 10 mg/d of prednisone or equivalent) may be approved after consultation with the study PI or Co-PI.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Patient with any prior immune related events (irAE) Grade 3 or higher that resulted in discontinuing or significant delay of dosing of immunotherapy
* Has received a live-virus vaccination within 30 days of planned treatment start.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial and Cervical Cancers
Enrollment: 50 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04-04 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 27 weeks
  Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rubinstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm